CLINICAL TRIAL: NCT05724121
Title: Observational Study of Cardiac Arrhythmias During Treatment With BTK Inhibitors or Venetoclax
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000923; 000923-H
Record Dates: First submitted 2023-02-10; First posted 2023-02-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11-26

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Waldenstr(SqrRoot)(Delta)m s Macroglobulinemia; Mantle Cell Lymphoma; Sudden Cardiac Death; Cardiac Arrhythmias; Hematologic Malignancies
Keywords: SUDDEN CARDIAC DEATH; Chronic Lymphocytic Leukemia (CLL); Ibrutinib Treatment; Atrial Fibrillation/Flutter; Ventricular Arrhythmias; Natural History
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Death, Sudden, Cardiac; Arrhythmias, Cardiac; Hematologic Neoplasms; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: includes all patients prior to starting therapy with a BTKi
- Cohort B: includes all patients already on therapy with a BTKi
- Cohort C: includes all patients prior to starting therapy with venetoclax

SUMMARY:
Background:

Bruton s tyrosine kinase inhibitors (BTKi) are used to treat a form of leukemia. But taking BTKi can also increase a person s risk of developing an abnormal heart rhythm. This can cause sudden death. In this natural history study, researchers want to learn how BTKi affects the heart.

Objective:

To identify and monitor the effects of BTKi on the heart.

Eligibility:

People aged 18 and older currently receiving or planning to receive BTKi or venetoclax.

Design:

Participants who have not yet started BTKi will have 2 required clinic visits: 1 before they start taking BTKi, and 1 about 6 months later. Participants who are already taking BTKi will have 1 required visit.

Participants will undergo multiple tests:

A physical exam, including collection of blood and saliva.

A test that measures heart activity via stickers placed on the chest.

A test that uses sound waves to capture images of the heart.

An exercise stress test that monitors heart activity and blood pressure while the participant works on a treadmill or stationary bike. Sound wave images of the heart may also be taken while the participant exercises.

Stress magnetic resonance imaging (MRI) may be done in place of an exercise test. Participants will lie on a table that slides into a tube. They will be given drugs to stress the heart while images are taken.

Participants may wear a device to monitor their heart at home.

Participants may have repeat visits if they develop heart symptoms or if they need to stop taking BTKi. They will have follow-up phone calls each year for up to 3 years.

DETAILED DESCRIPTION:
Study Description:

Pharmacologic therapy with BTK inhibitors (BTKi) is associated with an increased risk of cardiac arrhythmias which can lead to sudden death. There is currently no standard for cardiac screening or monitoring patients on BTKi. We hypothesize that thorough and routine comprehensive cardiac evaluations prior to starting therapy with BTKi and repeated during therapy with BTKi will result in earlier identification of cardiac arrhythmias with the goal of minimizing associated morbidity and mortality. In addition, venetoclax, a different standard therapy for chronic lymphocytic leukemia, has not been associated with increased cardiac adverse events and could serve as a control group.

Objectives:

Primary objective: Identify, monitor, and analyze the arrhythmogenic effects of BTKi as well as sudden death

Secondary objective: Assess the utility of different cardiac tests for identifying and monitoring cardiac arrhythmias in patients receiving BTKi or venetoclax

Exploratory objective: To examine the relationship between the development of cardiac arrhythmias in patients on BTKi as it relates to other variables

Endpoints:

Primary endpoint:

-A composite endpoint of clinically significant cardiac arrhythmias and sudden death in patients starting a BTKi (Cohort A) and in patients already receiving BTKi (Cohort B).

Secondary endpoints:

* Detection of arrhythmias on devices (rest/stress EKG, ambulatory EKG monitor, KardiaMobile)
* Arrhythmia (treatment emergent or worsening) in patients on BTKi
* Sudden death in patients on BTKi
* A composite endpoint of clinically significant cardiac arrhythmias and sudden death in patients starting venetoclax
* Difference in cardiac arrhythmias and sudden death between different BTKi groups (e.g., ibrutinib vs. non-ibrutinib group)
* Difference in cardiac arrhythmias and sudden death between BTKi and venetoclax groups

Exploratory endpoints:

* Pharmacokinetic levels of BTKi
* Duration of BTKi exposure
* Cumulative BTKi dose
* Genetic variants
* Cardiac structural remodeling
* Medical comorbidities
* Concomitant medications
* Substance use
* Identify risk factors or biomarkers for arrhythmia

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Currently receiving or planning to receive a BTKi or venetoclax.
2. Male or female, aged 18 or older
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any acute cardiac condition including myocardial infarction or decompensated heart failure within the past 3 months
2. Pregnancy or lactation- use of BTK inhibitors is contraindicated in pregnant or nursing individuals.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size of 135 subjects including men and women over 18 years old followed at the NIH Clinical Center who are either about to start a BTKi (Cohort A) or venetoclax (Cohort C) as well as those already taking BTKi (Cohort B)
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2027-04-08 (Estimated)

PRIMARY OUTCOMES:
arrhythmogenic cardiac effects of BTKi and sudden death within the first 12 months of BTKi therapy | 12 months
  1. Clinically significant cardiac arrhythmias while on a BTKi (treatment emergent in those without a history of arrhythmias and worsening of arrhythmia for those with an arrhythmia at the time of enrollment testing) within 12 months. For Cohort A, if a patient has an arrhythmia at the time of baseline testing, only worsening or new arrhythmias will be called an event. For Cohort B, all arrhythmias will be called an event. 2. Sudden death

SECONDARY OUTCOMES:
tests for identifying and monitoring cardiac arrhythmias in patients receiving BTKi | 36 months
  -Detection of arrhythmias on devices (rest EKG, stress EKG, ambulatory EKG monitor, KardiaMobile) -Clinically significant and other arrhythmias (treatment emergent or worsening) in patients on BTKi and on venetoclax -Sudden death -Composite endpoint of clinically significant cardiac arrhythmias and sudden death in patients starting venetoclax -Differences in cardiac arrhythmias and sudden death within BTKi (e.g., ibrutinib vs. non-ibrutinib group) -Differences in cardiac arrhythmias and sudden death between patients on BTKi and venetoclax

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Gruessner, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000923-H.html